CLINICAL TRIAL: NCT04414722
Title: Exploratory Pilot Studies to Demonstrate Mechanisms of Preventing Antibiotic-Associated Diarrhea and the Role for Probiotics
Brief Title: Mechanisms of Probiotics and Antibiotic-Associated Diarrhea
Acronym: OURBIOTIC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Maryland, Baltimore (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Daniel Merenstein, Director of Research Programs, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2020-2431; R33AT009622 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Antibiotic-associated Diarrhea
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Concurrent control yogurt and amoxicillin-clavulanate (Placebo Comparator): Yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12) and amoxicillin-clavulanate 875 mg-125 mg oral tablet, taken at the same time
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet; Other: Control Yogurt
- Control yogurt taken 4 hours after amoxicillin-clavulanate (Placebo Comparator): Yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12) taken 4 hours after amoxicillin-clavulanate 875 mg-125 mg oral tablet
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet; Other: Control Yogurt
- Concurrent BB-12 yogurt and amoxicillin-clavulanate (Active Comparator): Bifidobacterium animalis subsp. lactis BB-12-supplemented yogurt and amoxicillin-clavulanate 875 mg-125 mg oral tablet, taken at the same time
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet; Biological: BB-12
- BB-12 yogurt taken 4 hours after amoxicillin-clavulanate (Active Comparator): Bifidobacterium animalis subsp. lactis BB-12-supplemented yogurt taken 4 hours after amoxicillin-clavulanate 875 mg-125 mg oral tablet
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet; Biological: BB-12
- Amoxicillin-clavulanate (Other): Amoxicillin-clavulanate 875 mg-125 mg oral tablet
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet — Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet
  Other Names: Augmentin; Amoxicillin/clavulanic acid
Biological: BB-12 — Bifidobacterium animalis subsp. lactis BB-12 (BB-12)-supplemented yogurt
  Other Names: Bifidobacterium animalis subsp. lactis, BB-12
  Arms: BB-12 yogurt taken 4 hours after amoxicillin-clavulanate; Concurrent BB-12 yogurt and amoxicillin-clavulanate
Other: Control Yogurt — Yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12)
  Arms: Concurrent control yogurt and amoxicillin-clavulanate; Control yogurt taken 4 hours after amoxicillin-clavulanate

SUMMARY:
The focus of the study is to better understand the mechanisms causing antibiotic-associated diarrhea (AAD) and how probiotics may prevent some of the iatrogenic effects of antibiotic medications. One of the most common indications for probiotics is for prevention of antibiotic-associated diarrhea. Clinically, different probiotic strains have demonstrated the ability to prevent AAD; however, the mechanism of action behind this effect has not been elucidated. Data from several studies suggest that antibiotic-induced disruption of commensal bacteria in the colon results in a significant (up to 50%) reduction in short chain fatty acid (SCFA) production and a concomitant reduction in Na-dependent fluid absorption resulting in AAD. Probiotics have been shown to ameliorate a variety of gastrointestinal disease states and thus, the study investigators hypothesize that administration of a probiotic yogurt will protect against the development of AAD.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that, when administered in adequate amounts, confer a health benefit on the host. One of the most common indications for probiotic treatment is the prevention of antibiotic-associated diarrhea (AAD). Unfortunately, the efficacy of many probiotic products used for AAD is not supported by rigorous independent research, and non-evidence-based clinical usage is common. Data from several studies are consistent with the notion that antibiotic-induced disruption of commensal bacteria in the colon results in a significant reduction of short chain fatty acid (SCFA) production and a concomitant reduction in Na-dependent fluid absorption resulting in AAD. The probiotic strain being studied, Bifidobacterium animalis subsp. lactis BB-12 (BB-12), has been shown to ameliorate a variety of gastrointestinal disease states and is known to produce acetate at concentrations up to 50 mM in vitro. Thus, the investigators hypothesize that administration of BB-12 at the same time as antibiotic consumption will protect against the development of AAD through its ability to generate acetate directly, and also increase other SCFAs through cross-feeding of certain bacteria in the Firmicutes phylum such Clostridium, Eubacterium and Roseburia, which use acetate to produce butyrate.

The primary aim is to determine the ability of BB-12 to impact antibiotic-induced reduction in SCFA as reflected by the levels of acetate, the most abundant primary colonic SCFA, and assess temporal intervals of probiotic administration. The primary hypothesis is that antibiotics will result in a reduction in fecal SCFA, but BB-12 supplementation will protect against antibiotic-induced SCFA reduction and/or be associated with a more rapid return to baseline SCFA levels as compared to controls. Antibiotics also result in a decrease in total microbial counts and diversity in the gut microbiota, disrupting the homeostasis of the gut ecosystem and allowing colonization by pathogens. We hypothesize that concurrent administration of the probiotic and antibiotic is not necessary for the probiotic impact on SCFA.

The secondary aim will be to determine the ability of BB-12 to impact antibiotic-induced disruption of the gut microbiota with 16S ribosomal ribonucleic acid (rRNA) profiling, and assess temporal intervals of probiotic administration. The secondary hypothesis is that antibiotics will result in a decrease in the overall number and diversity of bacterial species present in the fecal microbiota, and further BB-12 supplementation will protect against antibiotic-induced shifts in the microbiota and/or will be associated with a more rapid return to a baseline microbiota composition as compared to controls. We hypothesize that concurrent administration of the probiotic and antibiotic is not necessary for the probiotic effect on the composition of the gut microbiota.

The tertiary aim is to longitudinally characterize the gut microbiota with high-throughput metatranscriptomics in order to generate complementary information on the impact of antibiotics plus and minus BB-12 on overall microbiome function. We hypothesize that acetate produced by BB-12 in situ will cross-feed butyrate producers in the Firmicutes phylum resulting in an up-regulation of butyrate biosynthetic pathways.

The long-term goal is to determine the impact of BB-12 on a variety of gastrointestinal disease states and ages, through high-level independent research. This mechanism elucidation is important for directing future translational and effectiveness research.

ELIGIBILITY:
Inclusion Criteria:

* Has the ability to read, speak, and write in English
* Has a refrigerator (for proper storage of the study yogurt)
* Has reliable telephone access
* Is between ages of 18-65 years
* Agree to refrain from eating yogurts, yogurt drinks, and other foods specified in the provided list
* Agree to collect stool samples and participate in follow-up calls as specified

Exclusion Criteria:

* Diabetes or asthma that requires medication
* Allergy to strawberry
* Active diarrhea (three or more loose stools per day for two consecutive days)
* Any gastrointestinal (or digestive tract) medications, i.e. medicines for irritable bowel syndrome, gastroesophageal (acid) reflux disease, inflammatory bowel disease, etc.
* History of heart disease, including valvulopathies or cardiac surgery, any implantable device or prosthetic
* History of gastrointestinal surgery or disease
* Lactose intolerance that prevents participant from eating yogurt
* Allergy to milk-protein
* Allergy to any component of the product or the yogurt vehicle
* Allergy to penicillin or cephalosporin class antibiotics
* Allergy to any of the following medications: a) Penicillin; b) Erythromycin; c) Tetracycline; d) Trimethoprim; e) Ciprofloxacin
* Women who are breastfeeding, pregnant, or planning to become pregnant during the study
* Was a participant in the "YOBIOTIC" study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, participants complete a 30-day run-in during which they refrain from probiotics and antibiotics. Participants who start/experience an exclusionary medication or nontransient health condition during run-in are withdrawn. Participants who take antibiotics during the run-in will delay the initiation of interventions until a full 30-day run-in cycle is complete. Participants who take non-study probiotics will document use and may continue with group assignment.
Groups:
- Concurrent Control Yogurt and Amoxicillin-clavulanate: Control yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12) and amoxicillin-clavulanate 875 mg-125 mg oral tablet, taken at the same time
- Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate: Control yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12) taken 4 hours after amoxicillin-clavulanate 875 mg-125 mg oral tablet
Period: Overall Study
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Started | 26 | 27 | 26 | 27 | 12
Completed | 17 | 18 | 19 | 20 | 8
Not Completed | 9 | 9 | 7 | 7 | 4
Not completed — Lost to Follow-up | 3 | 4 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 6 | 3 | 1 | 5 | 1
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 0
Not completed — Non-participatory | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate | Total
Number analyzed (Participants) | 26 | 27 | 26 | 27 | 12 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.15 (13.86) | 33.88 (14.79) | 30.18 (11.95) | 31.95 (14.09) | 26.30 (7.78) | 30.47 (2.998)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 14 | 17 | 5 | 71
  Male | 9 | 9 | 12 | 10 | 7 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 1 | 4 | 3 | 17
  Not Hispanic or Latino | 20 | 24 | 25 | 23 | 9 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 1 | 1 | 2 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 7 | 5 | 6 | 0 | 21
  White | 12 | 18 | 17 | 19 | 8 | 74
  More than one race | 5 | 1 | 0 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Levels of Fecal Short-chain Fatty Acid (With a Particular Focus on Acetate)
Description: Change from baseline levels of fecal short-chain fatty acid (with a particular focus on acetate)
Time Frame: day 7
Population: Participants were required to have baseline and Day 7 samples in order for this measurement to be taken.
  Participants that were not analyzed were missing a baseline or Day 7 comparator therefore were not analyzed.
Measure: Median (Inter-Quartile Range); unit: micromolar
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Number analyzed (Participants) | 12 | 13 | 11 | 14 | 6
micromolar | 23.55 [-51.55 to 78.8] | -13.9 [-30.1 to 24.7] | -19.5 [-41.1 to -8.3] | 7.25 [-51.2 to 31.1] | -21.7 [-34.6 to -4.0]

2. Primary Outcome: Change From Baseline Levels of Fecal Short-chain Fatty Acid (With a Particular Focus on Acetate)
Description: Change from baseline levels of fecal short-chain fatty acid (with a particular focus on acetate)
Time Frame: day 30
Population: Participants were required to have baseline and Day 30 samples in order for this measurement to be taken.
  Participants that were not analyzed were missing a baseline or Day 30 comparator therefore were not analyzed.
Measure: Median (Inter-Quartile Range); unit: micromolar
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Number analyzed (Participants) | 10 | 12 | 8 | 11 | 6
micromolar | 2.5 [-44.7 to 26.4] | 7.8 [-16.9 to 69.4] | 6.1 [-46.3 to 20.4] | -25.5 [-41.8 to 36.6] | -15.75 [-30.7 to 59.7]

3. Secondary Outcome: Percentage Change in Baseline Diversity of Bacterial Species in Fecal Microbiota
Description: Percentage Change in Baseline Diversity of Bacterial Species in Fecal Microbiota (based on the Shannon Diversity Index, percentage of change):
  This outcome measures the percentage change in baseline diversity of bacterial species in the fecal microbiota, using the Shannon Diversity Index. Percent change within each treatment group was calculated comparing the Shannon diversity index at each follow-up day (i.e., day 7) to day 0 (baseline). The Shannon Diversity Index is a commonly used method to quantify microbial diversity, incorporating both the richness (the number of different species) and evenness (the distribution of species) within a sample. A positive percentage change reflects an increase in microbial diversity, while a negative percentage change indicates a decrease in microbial diversity compared to the microbial diversity at baseline.
Time Frame: day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Number analyzed (Participants) | 17 | 12 | 17 | 18 | 7
percentage of change | -8.062 (17.52) | -8.994 (11.511) | -16.177 (16.053) | -13.479 (17.7) | -4.614 (9.691)

4. Secondary Outcome: Percentage Change in Baseline Diversity of Bacterial Species in Fecal Microbiota
Description: Percentage Change in Baseline Diversity of Bacterial Species in Fecal Microbiota (based on the Shannon Diversity Index, percentage of change):
  This outcome measures the percentage change in baseline diversity of bacterial species in the fecal microbiota, using the Shannon Diversity Index. Percent change within each treatment group was calculated comparing the Shannon diversity index at each follow-up day (i.e., day 14) to day 0 (baseline). The Shannon Diversity Index is a commonly used method to quantify microbial diversity, incorporating both the richness (the number of different species) and evenness (the distribution of species) within a sample. A positive percentage change reflects an increase in microbial diversity, while a negative percentage change indicates a decrease in microbial diversity compared to the microbial diversity at baseline.
Time Frame: day 14
Population: Participants were required to have baseline and Day 14 samples in order for this measurement to be taken.
  Participants that were not analyzed were missing a baseline or Day 14 comparator therefore were not analyzed.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Number analyzed (Participants) | 15 | 17 | 17 | 17 | 7
percentage of change | -1.456 (12.013) | -1.826 (10.395) | -5.999 (13.018) | -7.547 (10.808) | -2.374 (7.471)

5. Other Pre Specified Outcome: Change From Baseline Levels of Fecal Short-chain Fatty Acid (With a Particular Focus on Acetate)
Description: Change from baseline levels of fecal short-chain fatty acid (with a particular focus on acetate)
Time Frame: day 14
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: micromolar
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Number analyzed (Participants) | 11 | 12 | 11 | 14 | 6
micromolar | 1.6 [-24.5 to 66.3] | 0.6 [-10.1 to 63.0] | -37.8 [-53.0 to 23.6] | -13 [-36.6 to 29.9] | -5.3 [-31.2 to 23.1]

6. Other Pre Specified Outcome: Change From Baseline Levels of Fecal Short-chain Fatty Acid (With a Particular Focus on Acetate)
Description: Change from baseline levels of fecal short-chain fatty acid (with a particular focus on acetate)
Time Frame: day 21
Population: Participants were required to have baseline and Day 21 samples in order for this measurement to be taken.
  Participants that were not analyzed were missing a baseline or Day 21 comparator therefore were not analyzed.
Measure: Median (Inter-Quartile Range); unit: micromolar
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
Number analyzed (Participants) | 12 | 12 | 10 | 13 | 4
micromolar | -25.65 [-37.7 to 67.2] | -10.75 [-46.6 to 27.7] | -21.3 [-47.3 to -5.3] | -18.2 [-41.7 to 24.4] | -5.7 [-39.3 to 0.3]

ADVERSE EVENTS:
Time Frame: From baseline, through the 30-day run-in, and 30 days on-study (total 2 months)
Arm/Group | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Concurrent Control Yogurt and Amoxicillin-clavulanate | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate | Amoxicillin-clavulanate
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/26 | 0/27 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 1/26 | 0/27 | 0/12
Other Adverse Events (participants affected / at risk) | 14/26 | 18/27 | 17/26 | 15/27 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate (N=26) | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate (N=27) | Concurrent Control Yogurt and Amoxicillin-clavulanate (N=26) | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate (N=27) | Amoxicillin-clavulanate (N=12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent BB-12 Yogurt and Amoxicillin-clavulanate (N=26) | BB-12 Yogurt Taken 4 Hours After Amoxicillin-clavulanate (N=27) | Concurrent Control Yogurt and Amoxicillin-clavulanate (N=26) | Control Yogurt Taken 4 Hours After Amoxicillin-clavulanate (N=27) | Amoxicillin-clavulanate (N=12)
Loose stools (Gastrointestinal disorders) | 7 | 12 | 12 | 9 | 3
Flatulence (Gastrointestinal disorders) | 7 | 8 | 8 | 6 | 4
Stomach pain (Gastrointestinal disorders) | 5 | 8 | 5 | 6 | 2
Constipation (Gastrointestinal disorders) | 6 | 5 | 4 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 3 | 2 | 2
Fever (General disorders) | 0 | 2 | 1 | 0 | 0
Lack/loss of appetite (Gastrointestinal disorders) | 2 | 3 | 4 | 2 | 0
Rash (General disorders) | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 4 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Dryness of back of throat and tongue (General disorders) | 0 | 0 | 0 | 0 | 1
Cramps (General disorders) | 0 | 0 | 0 | 2 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT04414722/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT04414722/ICF_000.pdf